CLINICAL TRIAL: NCT06741631
Title: MyPEEPS LITE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); Northwestern University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Professor of Disease Prevention and Health Promotion and Professor of Population and Family Health; Associate Dean of Faculty Development, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAV4619; UH3AI169658 (NIH)
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): Participants randomized to the control arm will receive standard of care. This consists of HIV home testing every 6 months, information regarding sexual and other behaviors that potentiate one's risk for HIV infection, receipt of a fact sheet about PrEP and PEP, referrals to the local PrEP clinic, and referrals for local sexually transmitted disease testing.
- Intervention (Experimental): Participants randomized to the intervention arm will have access to MyPEEPS Mobile for the next 6 months. MyPEEPS Mobile is a secure web app with content delivered through games, scenarios, and role-plays within 22 mobile activities (true/ false questions, multiple choice, matching, videos).
  Interventions: Behavioral: MyPEEPS Mobile

INTERVENTIONS:
Behavioral: MyPEEPS Mobile — An evidence-based, digitally delivered mHealth sexual risk reduction intervention on HIV incidence.
  Arms: Intervention

SUMMARY:
This study will use community-informed advertisements and messages through electronic methods to recruit and retain a large (N=2,500), diverse national sample of high-risk young men who have sex with men (YMSM) and non-binary individuals that are assigned male sex at birth, 16-29 years of age to determine the efficacy of the MyPEEPS Mobile intervention on reduced incident HIV infections in comparison to a standard of care condition and to examine the degree to which reduced incident HIV infections occurs in the context of potential multilevel moderators and conceptual mediators. This is key to advancing HIV prevention among HIV-negative US persons at extremely high-risk for HIV seroconversion.

DETAILED DESCRIPTION:
In direct response to RFA-AI-21-018, Limited Interaction Targeted Epidemiology (LITE-2): To Advance HIV Prevention (UG3/UH3 Clinical Trial Optional), we proposed to harness innovative electronic methods to conduct a large, rigorous national study collecting and contextualizing epidemiological HIV incidence data in Young Men who have Sex with Men (YMSM) and testing the efficacy of MyPEEPS Mobile, an evidence-based, digitally delivered mHealth sexual risk reduction intervention on HIV incidence. We proposed to establish a large national cohort of 2,500 racially and ethnically diverse YMSM 16-29 years old, the age YMSM are most susceptible to HIV acquisition to identify theoretically-driven correlates of HIV seroconversion among a key population experiencing a disproportionate number of new HIV diagnoses.

Randomized controlled trials (RCTs) are considered the gold standard for estimating treatment efficacy because randomization mitigates risk of bias by balancing measured and unmeasured confounders across treatment groups. However, RCTs are costly, time-consuming, and can be challenging to conduct in certain context. We are therefore integrating the robust epidemiological data that we collected during the UG3 phase into the clinical trial design. That integration is a potentially appealing way to generate an external comparator cohort to increase the power of our RCT to estimate the effect of MyPEEPS Mobile on HIV incidence.

ELIGIBILITY:
Inclusion Criteria:

* Be between 16-29 years of age;
* Sex assigned at birth is male and identify gender as male or non-binary;
* Understand and read English;
* Live within US and its territories;
* Own or have access to a smartphone;
* Self-report anal sex with someone who has a penis in the last 12 months; and
* Be HIV-negative or status unknown

Exclusion Criteria:

* Individuals who identify as transgender

Ages: 16 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Sex assigned at birth is male and identify gender as male or non-binary
Enrollment: 2500 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
HIV Incidence | Baseline, 6 month follow up, 12 month follow up.
  OraQuick In-Home HIV Tests will be shipped to participants at baseline, 6 and 12 months.
Total Condomless Anal Sex Occurring in the Context of Insufficient PrEP Protection | Baseline, 6 month follow up, 12 month follow up.
  Condomless anal sex acts not protected by PrEP, defined as condomless anal sex acts in the prior 6 months without protection via PrEP. We will measure sexual risk with the AIDS-Risk Behavior Assessment.

SECONDARY OUTCOMES:
Self-Reported PrEP Initiation | Baseline, 6 month follow up, 12 month follow up.
  Self reported PrEP initiation variables will be measured for the purposes of characterizing the uptake of PrEP over the course of the study. We will use a self-reported approach to capture the date of initiation of medication, current use, and most recent date the medication was taken.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, Principal Investigator — Columbia University; Robert Garofalo, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Dustin Duncan, ScD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Columbia University, New York, New York